CLINICAL TRIAL: NCT02944877
Title: HOPE Social Media Intervention for HIV Testing and Studying Social Networks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, Los Angeles (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sean D Young, Associate Professor of Emergency Medicine and Informatics, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20205768; 1R01MH106415 (NIH)
Record Dates: First submitted 2016-02-05; First posted 2016-10-26 (Estimated); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: HIV

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): experimental
  Interventions: Behavioral: social media intervention
- control (Other): Other
  Interventions: Behavioral: social media intervention

INTERVENTIONS:
Behavioral: social media intervention — social media intervention

SUMMARY:
This study [HOPE: Harnessing Online Peer Education] seeks to determine the efficacy of using online social networks to scale peer community leader models to increase HIV prevention within African-American and Latino men who have sex with men. The peer community leader model, which teaches community popular opinion leaders about how to disseminate behavior changes messages throughout the community, has been proven to increase HIV prevention behaviors. Social media and online communities, such as Facebook, may be a cost-effective platform for scaling these models. Primarily upper middle-class White populations used the Internet in its early years, however, Internet use within African-American and Latino households has recently increased dramatically, especially on social media. People using the Internet may be at the highest risk for contracting HIV and are using novel Internet approaches to find sex partners, such as through social media. This is the first study to examine the effectiveness of the HOPE social media intervention to increase HIV testing among at-risk groups in the United States.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Male
* Sexually active with another man in the last 12 months
* Willing and capable of understanding and assenting to an online informed consent form
* Has (or willing to create) a social media page.

Exclusion Criteria:

* Does not satisfy inclusion criteria

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Young, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: experimental
  social media intervention: social media intervention with peer leaders for 12 weeks
- Control: Other
  social media intervention: social media intervention for 12 weeks without peer leaders
Period: Overall Study
Arm/Group | Intervention | Control
Started | 450 | 450
Completed | 421 | 418
Not Completed | 29 | 32

BASELINE CHARACTERISTICS:
Groups:
- Intervention: experimental
  social media intervention: social media intervention with peer leaders
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 450 | 450 | 900
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (9.8) | 31 (8.8) | 32 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 450 | 450 | 900
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White/European Descent | 39 | 28 | 67
  Race/Ethnicity: Latino/Caribbean | 301 | 319 | 620
  Race/Ethnicity: Black/African American | 72 | 73 | 145
  Race/Ethnicity: American Indian or Alaska Native | 8 | 7 | 15
  Race/Ethnicity: Asian or Pacific Islander | 18 | 16 | 34
  Race/Ethnicity: Other | 12 | 7 | 19
Region of Enrollment [Number; unit: participants]
  United States | 450 | 450 | 900

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Requesting HIV Self-Testing
Description: At home/self HIV testing kits can be requested to be ordered and will be provided to all participants who request it.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 450 | 450
Participants | 130 | 102

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/450 | 0/450
Serious Adverse Events (participants affected / at risk) | 0/450 | 0/450
Other Adverse Events (participants affected / at risk) | 0/450 | 0/450

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT02944877/Prot_SAP_000.pdf